CLINICAL TRIAL: NCT04128735
Title: The Prevalence of Diastolic Dysfunction in Morbidly Obese Patients Undergo Bariatric Surgery
Brief Title: Diastolic Dysfunction in Morbidly Obese Patients Undergo Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_2
Record Dates: First submitted 2019-04-02; First posted 2019-10-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Diastolic Dysfunction; Morbid Obesity
Keywords: Diastolic dysfunction; Morbid Obesity; Bariatric surgery
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Morbidly obese patients are at risk for diastolic cardiac dysfunction, which can lead to adverse event, such as, diastolic heart failure postoperatively. Preoperative screening by transthoracic echocardiogram is difficult due to anatomical challenge, therefore the prevalence of this problem may be underestimated. The investigator would like to perform transesophageal echocardiogram in this group of patients after anesthesia induction to demonstrate the true prevalence of this syndrome.

DETAILED DESCRIPTION:
Morbidly obese patients are at risk for both respiratory and cardiovascular abnormalities. Many cardiac problems were previously reported including left ventricular hypertrophy, right and left ventricular systolic dysfunction etc. Diastolic cardiac dysfunction can be found in normal left ventricular systolic function and can lead to diastolic heart failure postoperatively.

Preoperative screening by transthoracic echocardiogram is difficult due to anatomical challenge (thick chest wall, narrowing of inter-rib space), therefore the prevalence of this problem may be underestimated. Transesophageal echocardiogram provides better cardiac view, but requires sedation during procedure. So, it is not practical for out-patient setting. The investigator would like to perform transesophageal echocardiogram in this group of patients after anesthesia induction to demonstrate the true prevalence of this syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Every patient scheduled for bariatric surgery in Siriraj hospital

Exclusion Criteria:

* Patient refusal
* patient with contraindication for transesophageal echocardiogram such as preexisting esophageal disease, recent upper gastrointestinal bleeding, coagulopathy, etc. (according to American society of Echocardiography guideline)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Criteria for patient enrolled to bariatric surgery in Siriraj hospital
  * BMI more than 40 kg/m2
  * BMI more than 35 kg/m2 with hypertension, type 2 diabetes, hyperlipidemia, obstructive sleep apnea, chronic arthritis
  * age between 18 - 70 years old
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Prevalence of diastolic dysfunction | during surgery
  Prevalence of diastolic dysfunction according to American society of echocardiography definition

SECONDARY OUTCOMES:
Prevalence of other cardiac abnormalities | during surgery
  Number of patients with other cardiac abnormalities, both structural and functional abnormalities
Incidence of cardiac adverse events | within 24 hours after surgery
  Number of patients with cardiac adverse event: myocardial ischemia, pulmonary edema
Incidence of pulmonary adverse events | within 24 hours after surgery
  Number of patients experienced aspiration, desaturation, re-intubation
Incidence of oral and airway trauma | within 24 hours after surgery
  Number of patients with new loose teeth, sore throat, difficult to swallow, hoarseness of voice
Length of hospital stay | up to 5 days
  duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Aphichat Suphathamwit, M.D., Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cabrera Schulmeyer MC, Arriaza N. Good prognostic value of the intraoperative tissue Doppler-derived index E/e' after non-cardiac surgery. Minerva Anestesiol. 2012 Sep;78(9):1013-8. Epub 2012 Jun 14. PMID 22699700
- [Background] Hahn RT, Abraham T, Adams MS, Bruce CJ, Glas KE, Lang RM, Reeves ST, Shanewise JS, Siu SC, Stewart W, Picard MH. Guidelines for performing a comprehensive transesophageal echocardiographic examination: recommendations from the American Society of Echocardiography and the Society of Cardiovascular Anesthesiologists. J Am Soc Echocardiogr. 2013 Sep;26(9):921-64. doi: 10.1016/j.echo.2013.07.009. No abstract available. PMID 23998692
- [Result] Aljaroudi W, Alraies MC, Halley C, Rodriguez L, Grimm RA, Thomas JD, Jaber WA. Impact of progression of diastolic dysfunction on mortality in patients with normal ejection fraction. Circulation. 2012 Feb 14;125(6):782-8. doi: 10.1161/CIRCULATIONAHA.111.066423. Epub 2012 Jan 18. PMID 22261198